CLINICAL TRIAL: NCT03016689
Title: The Sinonasal Cavity as a Reservoir for Upper Airway Bacterial Development
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: MICRO-2016-25363
Record Dates: First submitted 2017-01-09; First posted 2017-01-10 (Estimated); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Oral and oropharyngeal swabs will be collected
Oversight: Data Monitoring Committee: No

SUMMARY:
While the maternal-newborn exchange of airway microbiota is well-documented, no studies have examined within-subject relationships among the mouth, sinuses, nasopharynx and lungs and the relative abundance of bacterial taxa at those sites. Recent evidence suggests the oral cavity may serve as a reservoir for pathogens that translocate to non-oral locations; oral-associated microbes infect most other body sites as evidence by 16S sequencing.

By using a combination of oral and throat swabs, together with nasal suction of mucus samples, the investigators will use metagenomic sequencing to characterize the composition of bacterial communities at each anatomical site. Beginning at birth, a time-series of swabs will be collected from each subject, and monitor changes in the development of microbiota over time. By doing so, our studies will illuminate airway trafficking of both beneficial and pathogenic microbes and may represent an essential pathophysiological step towards shifting the balance between airway health and disease.

DETAILED DESCRIPTION:
The study of microbial community dynamics is critically important to human health, including how to maintain or restore a healthy microbiome. Metagenomic studies have revolutionized microbiology by addressing these issues in a culture-independent manner, and have defined essential roles of the microbiota in host development. The initial development of gut microbiota begins in utero and is strongly influenced by exposures at birth (e.g. vaginal vs caesarean birth). The initial seeding by the mother's microflora and its ensuing bacterial succession is thought to have critical long-term impacts on human health. Recent longitudinal studies have documented a gradual increased in bacterial diversity, non-random community assembly, the effects of breast milk and introduction of table foods, and large taxonomic shifts as a result of antibiotics and environmental stresses that occur during infancy. Since perturbations of these early events have been linked to diabetes, cancer, mental health and a range of other maladies, efforts are underway to learn how manipulation of the infant microbiome to a "healthy" state translates into long-term clinical outcomes.

By contrast, little attention has been paid to factors that govern the early-life development of respiratory tract microbiota, including the oral cavity. At birth, the oral and nasopharyngeal flora resemble those of the maternal vaginal tract or skin (depending on mode of delivery). Preliminary datasets suggest that during the first year of life, the airway microbiome evolves into a rich, adult-like microbial ecosystem. The keystone colonizers of the airways are thought to condition the subsequent colonization by over 600 species, some of which serve to establish robust bacterial communities characteristic of human health. Other secondary colonizers are frequently implicated in oral and respiratory infections, including chronic sinusitis, pneumonia, and periodontal diseases. As an example, infant colonization by Streptococcus pneumoniae is an important risk factor for childhood middle ear disease. Early microbial communities, therefore, represent major factors that govern the colonization of the airways by both pathogenic and protective microbes during infant microbiome development. Understanding the acquisition of infant airway microbial communities and the factors that alter their composition is critical to the promotion of human health and the prevention of airway diseases that represent an annual multi-billion dollar burden on the US healthcare system.

While the maternal-newborn exchange of airway microbiota is well-documented, no studies have examined within-subject relationships among the mouth, sinuses, nasopharynx and lungs and the relative abundance of bacterial taxa at those sites. Recent evidence suggests the oral cavity may serve as a reservoir for pathogens that trans-locate to non-oral locations; oral-associated microbes infect most other body sites as evidence by 16S sequencing. However, two caveats make this bacterial metastasis controversial. First, that oral bacteria are not located solely in the mouth but are also found elsewhere in the airways makes their origin difficult to establish. Thus, the directionality of microbial exchange between airway niche spaces is not known. Secondly, most 16S ribosomal RNA (rRNA) surveys only reveal bacterial composition at the genus or phylum level, providing little information about strain lineages, and whether individual strains can migrate between sites. These data are critical to promote development of protective microbiota while restricting growth of recalcitrant pathogens.

A more complete understanding of this trafficking begins with in-depth, strain-level surveys of the bacterial communities present in each airway niche shortly after birth, and their development over time. As a step in this direction, this Academic Health Center-sponsored study will use metagenomic sequencing to assess the exchange of specific bacterial strains throughout the upper airways. Our mouse studies (explained elsewhere) will be complemented by a study of cystic fibrosis (CF) infants, who represent a unique population that facilitates the capture of oral, sinonasal, and lung microbiota over the first two years of life. By using a combination of oral and throat swabs, together with nasal suction of mucus samples, a metagenomic sequencing approach will be used to characterize the composition of bacterial communities at each anatomical site. Beginning at birth, the investigators will collect a time-series of swabs from each subject, and monitor changes in the development of microbiota over time. By doing so, our studies will illuminate airway trafficking of both beneficial and pathogenic microbes and may represent an essential pathophysiological step towards shifting the balance between airway health and disease.

EXPERIMENTAL PLAN The development of airway bacterial communities will be monitored in a small CF patient cohort. Since CF infants are monitored from birth and are routinely sampled for airway microbiota during routine outpatient visits as part of their standard-of-care, they represent a unique population to monitor bacterial trafficking between the oral, nasal and lung cavities. All newborns at the University of Minnesota (UMN) are genetically screened. Those testing positive for CF will be confirmed using a pilocarpine sweat test. Positive subjects (with 2 Cystic Fibrosis Transmembrane Conductance Regulator [CFTR] mutations) will then be sampled during the participants' visits to the CF treatment center; on average, infants will be seen every month for the first 6 months, every other month until 1 year of age, followed by quarterly visits to the UMN CF Center (in accordance with Cystic Fibrosis Foundation guidelines). As part of standard of care, nasal samples are collected by suction at each visit. Nylon swabs will also be used to sample each infant's buccal mucosa. Oropharyngeal swabs will also be obtained, which are considered to be an accurate proxy of lower airway (lung) microbiomes. Based on the number of CF newborns expected over the study period, the investigators plan to recruit up to 10 subjects. From each infant, up to 10 temporal swabs will be collected from each airway site (10 infants x 10 swabs x 3 sites = 300 samples). Swabs will be stored in saline, frozen at -80C and processed in parallel.

DNA will be extracted from each swab sample, and sequencing performed at the University of Minnesota Genomics Center.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF by sweat chloride test >60 mEq/L or by presence of two known CF genetic mutations
* Age 0-3 years
* Willingness to comply with study procedures
* Willingness of parent/guardian to provide written consent.

Exclusion Criteria:

• Presence of vasculitis or rheumatologic disorder

Ages: 7 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with Cystic Fibrosis who receive their care at the University of Minnesota Discovery Care Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The sinonasal cavity as a reservoir for upper airway bacterial development | 3 years
  The primary outcome measure will be the development and composition of bacterial communities throughout the respiratory tract during the first year of life. Community composition will be assessed using 16S rRNA sequencing, and differences between body sites will be calculated using standard ecological metrics.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hunter, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No